CLINICAL TRIAL: NCT03743194
Title: Pectoralis and Serratus Muscle Blocks for Analgesia After Minimally Invasive Cardiac Procedures
Brief Title: Pectoralis and Serratus Muscle Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-1125
Record Dates: First submitted 2018-10-31; First posted 2018-11-16 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Post Operative Pain Control
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupi HCl plus liposomal bupi (Active Comparator): Pectoral fascial plane or serratus anterior plane blocks (PECSII/SAP blocks) with bupivacaine HCl plus liposomal bupivacaine.
  An ultrasound guided pectoral fascial plane blocks (PECS I and II blocks) and Serratus anterior plane (SAP) block with injection of the local anesthetic.
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection; Drug: Placebo
- Control Group (Placebo Comparator): Standard parenteral analgesia technique with or without incisional local anesthetic infiltration: patients randomized to control group will be given parenteral opioids (such as fentanyl or hydromorphone) until they are converted to the enteral medications such as Percocet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exparel 266 MG Per 20 ML Injection — The local anesthetic (LA) used for the PECS II or serratus plane blocks will be a 0.5% bupivacaine HCL, not to exceed 2.5mg/kg or up to 150mg. The LA solution can be diluted with preservative free normal saline for smaller patients to allow for appropriate volume of injection. Treatment patients will also be given liposomal bupivacaine (EXPAREL, Pacira Pharmaceuticals, Inc. San Diego, CA) in a dose of 266 mg in 20 ml can be safely combined with bupivacaine HCL at a ratio not exceeding 2:1, but cannot be combined with other local anesthetics due to the concern of rapid release of encapsulated bupivacaine and subsequent local anesthetic toxicity.
  Other Names: Pectoralis and Serratus Muscle Blocks
  Arms: Bupi HCl plus liposomal bupi
Drug: Placebo — Patients randomized to standard analgesia technique will be given pain medications.
  Other Names: Standard analgesia technique (control, NO PECS /SAP blocks)

SUMMARY:
The overall research plan is PECS/SAP blocks with liposomal bupivacaine improve the Overall Benefit Analgesia Score averaged over the postoperative days 1, 2, and 3. A 20% reduction on geometric means (i.e., true ratio of geometric means of 0.80) in OBAS will be considered the minimal clinically important benefit.

DETAILED DESCRIPTION:
The primary aim is to determine whether a PECS/SAP block, using a mixture of bupivacaine and liposomal bupivacaine, provides superior recovery compared to routine parenteral and enteral analgesia in patients recovering from MICS. The primary outcome will be the simple multi-dimensional quality assessment, Overall Benefit Analgesia Score (OBAS score).53 Our secondary aims are to: 1) compare cumulative postoperative opioid consumption (pain medications administered over one-day periods quantified as morphine equivalents and provided by the EMR for the day of surgery and postoperative days 1, 2, and 3; 2) evaluate respiratory mechanics (forced expiratory volume in first minute (FEV1), forced vital capacity (FVC) and peak flow) after extubation on the postoperative days 1, 2 and 3 while patients remain hospitalized; and, (3) evaluate the Quality-of-Recovery-15 score on the postoperative days 1, 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years old;
2. Elective minimally invasive robotically-assisted mitral valve repair via anterolateral thoracotomy

Exclusion Criteria:

1. Weight less than 50 kg;
2. Pregnancy or lactation;
3. Emergency surgery and patients transferred from the ICU to the operating room;
4. Redo cardiothoracic surgery or post-operative reoperation within 72 hours of index procedure (including minor chest wall procedures including tube thoracostomy, thoracentesis or percutaneous drain placement);
5. Anticipated endotracheal intubation > 24 hours;
6. Anticipated non-study nerve block that provides analgesia to the intercostal nerves;
7. Active systemic or cardiopulmonary infection;
8. Mechanical circulatory support;
9. Allergy or contraindication to study local anesthetics;
10. Current chronic pain or routine opioid use (patients on chronic enteral opioids like Percocet or Vicodin) in a dose of > 30 mg of morphine-milligram-equivalents for at least 10 days in last 30 days;
11. Poorly controlled psychiatric disorders;
12. Clinically important current neurologic deficit;
13. Active liver disease or cirrhosis;
14. Pacemaker generator or breast implants ipsilateral to surgery;
15. Previous participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Alfirevic, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Alfirevic A, Marciniak D, Duncan AE, Kelava M, Yalcin EK, Hamadnalla H, Pu X, Sessler DI, Bauer A, Hargrave J, Bustamante S, Gillinov M, Wierup P, Burns DJP, Lam L, Turan A. Serratus anterior and pectoralis plane blocks for robotically assisted mitral valve repair: a randomised clinical trial. Br J Anaesth. 2023 Jun;130(6):786-794. doi: 10.1016/j.bja.2023.02.038. Epub 2023 Apr 11. PMID 37055276

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine HCl plus liposomal bupivacaine: The treatment group received Pectoral fascial plane or serratus anterior plane blocks (PECSII/SAP blocks) with bupivacaine HCl plus liposomal bupivacaine.
  An ultrasound guided pectoral fascial plane blocks (PECS I and II blocks) and Serratus anterior plane (SAP) block with injection of the local anesthetic.
  Exparel 266 MG Per 20 ML Injection: The local anesthetic (LA) used for the PECS II or serratus plane blocks will be a 0.5% bupivacaine HCL, not to exceed 2.5mg/kg or up to 150mg. The LA solution can be diluted with preservative free normal saline for smaller patients to allow for appropriate volume of injection. Treatment patients will also be given liposomal bupivacaine (EXPAREL, Pacira Pharmaceuticals, Inc. San Diego, CA) in a dose of 266 mg in 20 ml can be safely combined with bupivacaine HCL at a ratio not exceeding 2:1, but cannot be combined with other local anesthetics due to the concern of rapid release of encapsulated bupivacaine and subsequent local anesthetic toxicity.
  Placebo: Patients randomized to standard analgesia technique will be given pain medications.
Period: Overall Study
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
Started | 105 | 105
Completed | 98 | 96
Not Completed | 7 | 9
Not completed — Protocol Violation | 7 | 7
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 56 (11) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 74 | 80 | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 92 | 88 | 180
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 3 | 3
ASA status [Count of Participants; unit: Participants] — The ASA Physical Status Classification System has been in use for over 60 years. The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. The classification system alone does not predict the perioperative risks, but used with other factors (eg, type of surgery, frailty, level of deconditioning), it can be helpful in predicting perioperative risks. ASA takes values from I to VI, representing from a normal healthy patient to a declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    III | 79 | 79 | 158
    IV | 19 | 17 | 36
Smoking status [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 5
  No | 77 | 78 | 155
  Former | 19 | 15 | 34
Coronary arterial disease [Count of Participants; unit: Participants] | 6 | 3 | 9
Hypertension [Count of Participants; unit: Participants] | 31 | 27 | 58
Previous myocardial infarction [Count of Participants; unit: Participants] | 2 | 0 | 2
Previous vascular disease [Count of Participants; unit: Participants] | 1 | 0 | 1
Cerebrovascular disease [Count of Participants; unit: Participants] | 0 | 0 | 0
Diabetes mellitus [Count of Participants; unit: Participants] | 1 | 2 | 3
Renal failure [Count of Participants; unit: Participants] | 0 | 0 | 0
Left ventricular EF (% of ejection fraction) [Median (Inter-Quartile Range); unit: %of blood pumped out from left ventricle] — Ejection fraction is measured as a percentage of the total amount of blood in your heart that is pumped out with each heartbeat
  %of blood pumped out from left ventricle | 63 [60 to 67] | 61 [58 to 66] | 62 [60 to 66]
Baseline peak flow [Mean (Standard Deviation); unit: L/s] | 7.3 (2.7) | 7.4 (2.3) | 7.3 (2.5)
Baseline FEV1 [Mean (Standard Deviation); unit: L] — Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. Higher values suggests better lung function.
  L | 3.2 (0.8) | 3.3 (0.7) | 3.2 (0.7)
Baseline FVC [Mean (Standard Deviation); unit: L] — Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible. Higher values indicate better lung function.
  L | 4.1 (1.0) | 4.2 (0.9) | 4.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Overall Benefit Analgesia Score
Description: Our primary outcome, Overall Benefit Analgesia Score (OBAS), was measured daily by investigators blinded to treatment on postoperative Days 1 to 3.Potential scores of the seven-item questionnaire ranged from 0 to 28 points. Higher scores means worse conditions.
Time Frame: Postoperative day 1-3
Population: Some were some missing on each groups at each day during POD1- POD3. But since the statistical analysis used mixed model thus it could deal with missing as long as patients were not completely missing on all postoperative 3 days. Only 1 patient was missing on all postoperative 3 days, his outcome was imputed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
Number analyzed (Participants) | 98 | 96
score on a scale
  POD 1: number analyzed (Participants) | 96 | 94
  POD 1 | 4 [2 to 7] | 5 [2 to 6]
  POD 2: number analyzed (Participants) | 96 | 93
  POD 2 | 3 [2 to 6] | 3 [2 to 5]
  POD 3: number analyzed (Participants) | 93 | 92
  POD 3 | 2 [1 to 4] | 2 [1 to 4]
Statistical Analysis 1: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; A mixed effects linear model with repeated measures assuming an auto-regressive correlation structure was used to estimate the ratio of geometric means (treatment vs control). One patient from the control group whose measurements were all missing was conservatively imputed to have total OBAS of 2, 1, and 0 at postoperative Days 1, 2, and 3, respectively, assuming the best observed outcome for any control patient at that time. Total OBAS score was log transformed; Test type: Superiority; p = 0.75, Linear mixed model; Geometric mean ratio = 0.98, 95% CI 2-sided [0.85 to 1.13]
Statistical Analysis 2: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; A complete-case analysis (assumed that one patient was missing at random) was conducted as a sensitivity analysis. The ratio of geometric means (treatment vs control) was estimated using a mixed effects linear model with repeated measures assuming an auto-regressive AR(1) correlation structure; Test type: Superiority; p = 0.71, linear mixed model; Geometric mean ratio = 0.97, 95% CI 2-sided [0.83 to 1.14]
Statistical Analysis 3: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; The total OBAS was averaged over 3 postoperative days for the sensitivity analysis. A Wilcoxon rank-sum test with Hodges-Lehmann estimation was used to estimate the median of differences (each OBAS in the treatment group was compared with each OBAS in the control group to calculate the difference); Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.08, 95% CI 2-sided [-0.5 to 0.67]

2. Secondary Outcome: Cumulative Opioid Consumption Over Postoperative 3 Days
Description: Cumulative 72-hour postoperative opioid consumption (mg IV morphine equivalents)
Time Frame: 72 hours postoperative
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
Number analyzed (Participants) | 98 | 96
mg morphine equivalents | 118 [53 to 190] | 113 [53 to 188]
Statistical Analysis 1: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; Test type: Superiority — The ratio of geometric means was estimated through a generalized linear model with log transformed cumulative opioid consumption as the outcome and treatment group as the exposure. A multiple testing adjustment was applied (0.05/4 = 0.0125), thus 98.75% CI was provided; p = 0.94, Regression, Linear; Geometric mean ratio = 1.01, 98.75% CI 2-sided [0.73 to 1.40]

3. Secondary Outcome: Postoperative FEV1
Description: Pulmonary Mechanics measure: The FEV1 (forced expiratory volume in 1 seconds) in litters, measured using Easy on-PC Spirometry System (ndd Medical, Andover MA) with the patient in the sitting position. Measurements will be done on postoperative mornings 1, 2 and 3. The average of 3 days measurement will be calculated.
Time Frame: Postoperatively day 1 -3
Population: Some patients were missing on some measurements during POD1-POD3.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
Number analyzed (Participants) | 98 | 96
L
  POD1: number analyzed (Participants) | 76 | 66
  POD1 | 1.3 (0.4) | 1.3 (0.4)
  POD2: number analyzed (Participants) | 75 | 85
  POD2 | 1.4 (0.6) | 1.4 (0.5)
  POD3: number analyzed (Participants) | 78 | 82
  POD3 | 1.6 (0.6) | 1.6 (0.6)
Statistical Analysis 1: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; The difference in means was estimated through a mixed effects linear model with repeated measures assuming an auto-regressive correlation structure. Treatment effect was reported each day separately due to significant time-treatment interaction; Test type: Superiority — Difference in means at POD1; p = 0.36, Linear mixed model; Mean Difference (Final Values) = 0.08, 99.6% CI 2-sided [-0.17 to 0.32]
Statistical Analysis 2: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Difference in mean at POD2; p = 0.79, Linear mixed model; Mean Difference (Final Values) = -0.02, 99.6% CI 2-sided [-0.26 to 0.22]
Statistical Analysis 3: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Difference in mean at POD3; p = 0.39, Linear mixed model; Mean Difference (Final Values) = -0.07, 99.6% CI 2-sided [-0.31 to 0.17]

4. Secondary Outcome: Postoperative FVC
Description: Pulmonary Mechanics measure: the FVC (Forced Vital Capacity) in litters will be measured using Easy on-PC Spirometry System (ndd Medical, Andover MA) with the patient in the sitting position. Measurements will be done on postoperative mornings 1, 2 and 3. The average of 3 days measurement will be calculated.
Time Frame: Postoperative day 1 -3
Population: Some patients were missing on measurements during POD 1-POD3.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
Number analyzed (Participants) | 98 | 96
L
  POD1: number analyzed (Participants) | 76 | 66
  POD1 | 1.7 (0.6) | 1.7 (0.6)
  POD2: number analyzed (Participants) | 75 | 85
  POD2 | 1.8 (0.8) | 1.9 (0.7)
  POD3: number analyzed (Participants) | 80 | 82
  POD3 | 2.1 (0.8) | 2.2 (0.8)
Statistical Analysis 1: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Difference in mean in POD1; p = 0.51, Linear mixed model; Mean Difference (Final Values) = 0.07, 99.6% CI 2-sided [-0.25 to 0.4]
Statistical Analysis 2: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.91, Linear mixed model — Mean difference at POD2; Mean Difference (Final Values) = -0.01, 99.6% CI 2-sided [-0.33 to 0.30]
Statistical Analysis 3: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Difference in mean at POD3; p = 0.31, Linear mixed model; Mean Difference (Final Values) = -0.11, 99.6% CI 2-sided [-0.43 to 0.21]

5. Secondary Outcome: Postoperative Peak Flow
Description: Pulmonary Mechanics measure: the peak flow (peak expiratory flow) in litters per second will be measured using Easy on-PC Spirometry System (ndd Medical, Andover MA) with the patient in the sitting position. Measurements will be done on postoperative mornings 1, 2 and 3. The average of 3 days measurement will be calculated.
Time Frame: Postoperative day 1-3
Population: Some patients were missing on some measurements during POD1-POD3.
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
Number analyzed (Participants) | 98 | 96
L/s
  POD1: number analyzed (Participants) | 76 | 66
  POD1 | 3.1 (1.5) | 3.0 (1.2)
  POD2: number analyzed (Participants) | 75 | 85
  POD2 | 3.2 (1.5) | 3.2 (1.3)
  POD3: number analyzed (Participants) | 80 | 82
  POD3 | 3.4 (1.7) | 3.6 (1.7)
Statistical Analysis 1: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Difference in means at POD1; p = 0.36, Linear mixed model; Mean Difference (Final Values) = 0.22, 99.6% CI 2-sided [-0.47 to 0.91]
Statistical Analysis 2: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.97, Linear mixed model; Mean Difference (Final Values) = 0.01, 99.6% CI 2-sided [-0.66 to 0.67]
Statistical Analysis 3: Comparison: Bupivacaine HCl plus liposomal bupivacaine vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Difference in means at POD3; p = 0.36, Linear mixed model; Mean Difference (Final Values) = -0.21, 99.6% CI 2-sided [-0.88 to 0.46]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Bupivacaine HCl plus liposomal bupivacaine | Control Group
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/96
Other Adverse Events (participants affected / at risk) | 0/98 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT03743194/Prot_SAP_000.pdf